CLINICAL TRIAL: NCT03183336
Title: Horizontal Ridge Augmentation of the Mandible Using Interpositional Autogenous Block Grafts Versus Onlay Block Grafts; Randomized Controlled Clinical Trial
Brief Title: Horizontal Ridge Augmentation of the Mandible Autogenous Block Grafts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed H Osman, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cebc.cairou
Record Dates: First submitted 2017-06-06; First posted 2017-06-12 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Horizontal Ridge Deficiency; Block Graft

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interpositional block graft (Experimental): ridge split interpositional block graft
  Interventions: Procedure: ridge split interpositional block graft
- Onlay block graft (Active Comparator): decortication onlay block graft
  Interventions: Procedure: decortication Onlay block graft

INTERVENTIONS:
Procedure: ridge split interpositional block graft
  Arms: Interpositional block graft
Procedure: decortication Onlay block graft
  Arms: Onlay block graft

SUMMARY:
20 subjects presenting with horizontal mandibular ridge width less than 5 mm were selected and randomly divided two groups (10 in each group). the first group received interpositional block grafts (harvested from the chin and ramus) covered with Platelet-rich fibrin membrane. the second group received onlay block grafts (harvested from the chin and ramus) and covered with Platelet-rich fibrin membrane. the grafts are left for 4 months. the alveolar ridge width dimensions is then measured using radiographic analysis using cone-beam computed tomography scans

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with a minimum vertical bone height above the inferior alveolar canal of 10mm in the edentulous region.

Patients should have ridge thickness less than 5mm measured 2mm from the alveolar crest Patients should be free from any systemic disease that may affect normal healing of bone, and predictable outcome.

Exclusion Criteria:

* Patients with any systemic disease that may affect normal bone healing. Patients with drug allergies, drug or alcohol abuse, periodontal diseases or poor oral hygiene

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
alveolar ridge width gained | 4 months
  radiographic analysis following ridge augmentation using Cone beam computed tomography

SECONDARY OUTCOMES:
patient morbidity following the surgical procedure | 14 days
  pain value on pain scale

IPD SHARING:
Plan to Share IPD: Yes